CLINICAL TRIAL: NCT02036996
Title: Official Title Evaluation of EarlySense; a Contact-less Heart and Respiration Rate Monitoring in Sleep Lap Examined Evaluation of EarlySense; a Contact-less Heart and Respiration Rate Monitoring in Sleep Lap Examined
Brief Title: Evaluation of EarlySense; a Contact-less Heart and Respiration Rate Monitoring in Sleep Lap Examined
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ES-CLC-2013_Prot_4
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Over Weight; Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to collect heart rate, respiration data and motion data of patients admitted to sleep lab and to determine the current accuracy level of the EarlySense system vs. the standard system, and predicate device for EarlySense (Embla) used in sleep lab in monitoring heart rate and respiration rates monitors (ECG, respiratory belts, oximeter) that are currently used in the sleep lab among different population (Obese, patients with or without apnea, patients with or without arrhythmia). It is emphasized that no interpretations or clinical decisions will be made based on data received from the ES study device.

DETAILED DESCRIPTION:
The study objective is to collect heart rate, respiration rate and motion data of patients admitted to sleep lab and to determine the accuracy level of the EarlySense system vs. the monitors used in sleep lab (e.g., Polysomnography, respiratory belts, ECG, etc..) . Data regarding sleep condition, scoring and quality of sleep and in and out of bed status, patient turns will also be collected and compared to data collected by EarlySense contactless monitor. Different patient population will be monitored including obese, morbidly obese, patients with or without obstructive/central apnea, patients with or without arrhythmia as well as healthy population who arrive to sleep lab for general evaluation will be monitored

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years or more 2. Is willing to sign the consent form.

Exclusion Criteria:

* Age < 18 years
* Is not willing to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Different patient population will be monitored including obese, morbidly obese, patients with or without apnea, patients with or without arrhythmia as well as healthy population who arrive to sleep lab for general evaluation will be monitored
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Determine the detection rate and the accuracy of the EarlySense system in measuring HR and RR and motion as well as capability of system to detect patient turns, bed-exit and entries | one year
  Determine the detection rate and the accuracy of the EarlySense system in measuring HR and RR and motion as well as capability of system to detect patient turns, bed-exit and entries

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, Prof., Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel